CLINICAL TRIAL: NCT02866747
Title: A Phase I/II Multicenter Trial Evaluating the Association of Hypofractionated Stereotactic Radiation Therapy and the Anti-Programmed Death-ligand 1 (PD-L1) Durvalumab (Medi4736) for Patients With Recurrent Glioblastoma (STERIMGLI)
Brief Title: A Study Evaluating the Association of Hypofractionated Stereotactic Radiation Therapy and Durvalumab for Patients With Recurrent Glioblastoma
Acronym: STERIMGLI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16TETE04
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Arm A: radiation therapy alone (Active Comparator): Hypofractionated stereotactic radiation therapy (hFSRT) 24 Gray (Gy), 8 Gy per fraction preferentially at 80% isodose (60 to 90 % accepted), 3 fractions scheduled on Day 1 of the radiotherapy (RT), Day 3 RT and Day 5 RT.
  Interventions: Radiation: Hypofractionated stereotactic radiation therapy
- Arm B: combined treatment (Experimental): hFSRT 24 Gy, 8 Gy per fraction preferentially at 80% isodose (60 to 90 % accepted), 3 fractions scheduled on Day 1 RT, Day 3 RT and Day 5 RT, combined with Durvalumab infusion: first administration of Durvalumab* on Day 5 RT (i.e. the same day after the last fraction of radiation, corresponding to the Day 1 for Durvalumab treatment) and then administration of Durvalumab 1500 milligrams (mg) every four weeks.
  * Dosing 750 mg or 1500 mg, according to the recommended combination schema determined in phase I.
  Interventions: Radiation: Hypofractionated stereotactic radiation therapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Hypofractionated stereotactic radiation therapy
Drug: Durvalumab
  Arms: Arm B: combined treatment

SUMMARY:
This study is a phase I/II, national, multicenter, open-label study starting with a Phase I part followed by a Phase II part.

The phase I part of the study aims to evaluate the safety of the association of hypofractionated stereotactic radiation therapy (hFSRT) and the anti-PD-L1 Durvalumab immunotherapy in patients with recurrent glioblastoma. A maximum number of 12 patients will be enrolled in this phase I part.

Once the recommended combination schema will be declared, patients will be enrolled in the Phase II part of the study in order to evaluate the efficacy (overall survival) of the combined treatment in recurrent glioblastoma. In this Phase II part, 100 patients will be assigned by randomization to one of the two following arms:

* Arm A (control arm): Radiation therapy alone
* Arm B (Experimental arm): Combined treatment with Anti-PD-L1 Durvalumab

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at time of study entry.
2. Previous histopathologic confirmation of glioblastoma.
3. Any line of recurrence of glioblastoma proven by contrast enhanced MRI within 28 days prior to the first fraction of RT, per modified RANO criteria (Wen et al JCO 2010).

   Note: Recurrence is defined as progression following therapy (i.e., chemotherapy, radiation, second surgery).
4. Recurrent nodule of an histologically confirmed diagnosis of World Health Organization (WHO) Grade IV malignant glioma (Glioblastoma) occurring in or out the previous irradiation fields.
5. Recurrent disease documented by MRI evidence with a size of the recurrence evaluated on T1 post-gadolinium sequence ≤35mm.
6. Patient for which a re-irradiation (by hFSRT) has been decided by the multidisciplinary medical board.
7. Patients with measurable disease.
8. Prior radiotherapy must be ended at least 12 weeks before the first fraction of RT (unless progressive disease outside of the radiation field or histopathologic confirmation of unequivocal tumor to eliminate pseudoprogression images according to RANO recommendations, Wen et al JCO 2010).
9. In case of previous anti-VEGF/VEGFR targeted therapy: at least 28 days between the last injection of anti-VEGF/VEGFR targeted therapy and the first fraction of RT.
10. Karnofsky performance status ≥70.
11. Adequate hematologic, renal and hepatic function, as defined below:

    * Absolute Neutrophil Count ≥ 1500/mm3
    * Haemoglobin ≥ 9.0 g/dL
    * Platelet count ≥ 100,000/mm3
    * Total bilirubin ≤ 1.5 x ULN (for patient with confirmed Gilbert's syndrome,
    * Total bilirubin ≤ 3 x ULN)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
    * Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min, using the Cockcroft-Gault formula:

      * Female CrCl = (140 - age in years) x weight in kg x 0.85 /72 x serum creatinine in mg/dL
      * Male CrCl = (140 - age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL
12. Female Patients must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥ 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
13. Written informed consent and any locally required authorization (e.g., Social security for France (Health Insurance)) obtained from the patient prior performing any protocol-related procedures, including screening evaluations.
14. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Multifocal GBM recurrence (exception: multisite nodular recurrence (maximum: 2 sites) that can be irradiated by hFSRT according to investigator's judgement).
2. Distance between tumor and optic ways including chiasma or brainstem <1 cm.
3. Prior re-irradiation (except if fulfilling the following requirements: ended at least 6 months before the first fraction of RT in the study, localized outside the target of interest for the trial, and previously re-irradiated lesion controlled at the time of study entry).
4. Prior exposure to Durvalumab or other anti-PD-1, anti-PD-L1, anti-CTLA4 antibodies.
5. Patient who received a live vaccine within 30 days prior to the first fraction of RT.
6. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within 28 days prior to the first fraction of RT.
7. Current or prior use of immunosuppressive medication within 10 days before the first fraction of RT (exception: systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent are allowed as well as steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) - Topical, inhaled, nasal and ophthalmic steroids are not prohibited).
8. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
9. Presence of diffuse leptomeningeal disease or extracranial disease.
10. Active suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener's granulomatosis and Hashimoto's thyroiditis).

    Note: participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger, are permitted to enroll.
11. Known primary immunodeficiency or active HIV.
12. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months indicated by positive test for hepatitis B surface antigen (HBV sAG) or hepatitis C virus antibody.
13. History of organ transplant requiring use of immunosuppressive medication.
14. History of active tuberculosis.
15. Current pneumonitis or interstitial lung disease.
16. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses.
17. Other invasive malignancy within 2 years prior to entry into the study, except for those treated with surgical therapy only.
18. History of severe allergic reactions to any unknown allergens or any components of the study drug.
19. Any prior Grade ≥ 3 immune-related adverse event (irAE) or any prior corticosteroid-refractory irAE.
20. Participation in any other clinical trial involving another investigational product within 4 weeks prior to the first fraction of RT.
21. Participation in any other clinical trial which delivered a dose >60 Gy for the primo-treatment for glioblastoma.
22. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing highly effective method of birth control.
23. Any condition that, in the clinical judgment of the investigator, is likely to prevent the patient from complying with any aspect of the protocol or that may put the patient at unacceptable risk.
24. Mental impairment (psychiatric illness/social situations) that may compromise the ability of the patient to give informed consent and comply with the requirements of the study.
25. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose Limiting Toxicities (DLT) incidence | 8 months
  For each patient of the phase I part, DLT incidence will be evaluated until one month after the last radiotherapy fraction.
Phase II: overall survival | 36 months post randomization

SECONDARY OUTCOMES:
Phase I and II: Intracranial progression-free interval | 27 months
  Intracranial progression-free interval is defined by the time from inclusion (for phase I) or randomization (for phase II) to local or distant (outside the re-irradiated volume) progression. Patients without progression at last follow-up news are censored at this date.
Phase I: Safety and tolerability according to the classification of the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.03 | 19 months
Phase I and II: Quality of life using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ C30). | 27 months
Phase I and II : Quality of life using the using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Brain Neoplasm (QLQ-BN20). | 27 months
Phase I and II: Neurologic and neurocognitive functions using Neurologic Assessment in Neuro-Oncology (NANO) scale. | 27 months
Phase I and II: Neurologic and neurocognitive functions using Neurologic Assessment in Montreal Cognitive Assessment (MoCA) tests. | 27 months
Phase II: Time to Quality of Life (QoL) deterioration. | 27 months
  Time to QoL deterioration is defined as the time interval between randomization and first decrease in QoL score greater or equal to 5 points. Patients without such a QoL decrease will be censored at last follow-up news or at initiation of a new therapeutic strategy.
Phase II: time to neurocognitive deterioration | 27 months
  Time to neurocognitive deterioration is defined as the time interval between randomization and first of 3 points difference in MoCA as minimal clinically important difference. Patients without such a neurocognitive decrease will be censored at last follow-up news or at initiation of a new therapeutic strategy.
Phase II: Immune-related intracranial progression-free interval | 27 months
  Immune-related intracranial progression-free interval is defined by the time from randomization to local or distant (outside the re-irradiated volume) progression (based on immunotherapy Response Assessment for Neuro-Oncology iRANO). Patients without progression at last follow-up news are censored at this date.
Phase II: Acute and late toxicities according to the classification of the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) version 4.03 | 27 months

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut de Cancerologie de L'Ouest, Angers
  - Hopital Avicenne, Bobigny
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Institut Regional Du Cancer de Montpellier, Montpellier
  - Hopital Pitie Salpetriere, Paris
  - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pouessel D, Ken S, Gouaze-Andersson V, Piram L, Mervoyer A, Larrieu-Ciron D, Cabarrou B, Lusque A, Robert M, Frenel JS, Uro-Coste E, Olivier P, Mounier M, Sabatini U, Sanchez EH, Zouitine M, Berjaoui A, Cohen-Jonathan Moyal E. Hypofractionated Stereotactic Re-irradiation and Anti-PDL1 Durvalumab Combination in Recurrent Glioblastoma: STERIMGLI Phase I Results. Oncologist. 2023 Sep 7;28(9):825-e817. doi: 10.1093/oncolo/oyad095. PMID 37196069